CLINICAL TRIAL: NCT05006586
Title: Rectovaginal Fistula Repair Predictors of Outcome and Results After Surgical Management
Brief Title: Rectovaginal Fistula Repair
Status: Completed | Type: Observational
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Other Study IDs: RVF - quality of life
Record Dates: First submitted 2021-06-14; First posted 2021-08-16 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Fistula Vagina; Fistula;Rectal
Keywords: Rectovaginal fistula; Surgical repair; Quality-of-life
MeSH Terms: conditions — Vaginal Fistula; Rectal Fistula; Rectovaginal Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- RVF: All patients having undergone repair for rectovaginal fistula

SUMMARY:
This study is a prospective evaluation of quality-of-life after rectovaginal fistula repair at our institution

DETAILED DESCRIPTION:
All patient having undergone rectovaginal fistula repair at Uppsala University Hospital 2003-2018. An invitation to join the study was sent to all patients. Those who answered were then sent Rand 36/SF36 questionnaire as a follow-up together with some general questions concerning whether the rectovaginal fistula was healed or not.

ELIGIBILITY:
Inclusion Criteria:

* Undergone RVF repair at Uppsala University Hospital 2003-2018

Exclusion Criteria:

* Fistula due to gender reconstructive surgery

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women undergoing RVF repair att Uppsala University Hospital. A quality-of-life follow-up is planned.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
Surgical repair | Assessed on average 3 months postoperatively
  Rate of fistula closure

SECONDARY OUTCOMES:
Health-related Quality-of-life | Through study completion, on average 10 years
  SF36 questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Akademiska Sjukhuset (Uppsala University hospital), Uppsala, Sweden

REFERENCES:
- [Derived] Soderqvist EV, Cashin PH, Graf W. Surgical treatment of rectovaginal fistula-predictors of outcome and effects on quality of life. Int J Colorectal Dis. 2022 Jul;37(7):1699-1707. doi: 10.1007/s00384-022-04206-7. Epub 2022 Jul 2. PMID 35779081